CLINICAL TRIAL: NCT05479656
Title: A Better Trunk and Lower Limb Control for a Better Mobility: Assessment of a Re-entrainment Program in Autosomal Recessive Spastic Ataxia of Charlevoix-Saguenay
Brief Title: A Rehabilitation Program to Increase Balance and Mobility in Ataxia of Charlevoix-Saguenay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Élise Duchesne (Other)
Collaborators: Muscular Dystrophy Canada (Other)
Responsible Party: Sponsor-Investigator, Élise Duchesne, Professor, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-010
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Autosomal Recessive Spastic Ataxia of Charlevoix-Saguenay
MeSH Terms: conditions — Spastic ataxia Charlevoix-Saguenay type

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training program (Experimental): 8-week rehabilitation program aimed at increasing trunk and lower limb motor control on balance and walking abilities, and accomplishment of activities of daily living.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — 8-week rehabilitation program aimed at increasing trunk and lower limb motor control on balance and walking abilities, and accomplishment of activities of daily living.

SUMMARY:
This exploratory study used a pre-post test design. The supervised rehabilitation program was performed three times a week for 8 weeks (two sessions at a rehabilitation gym and one pool session). Outcome measures included Ottawa sitting scale, 30-Second Chair Stand test, Berg Balance Scale, 10-Meter Walk Test, 6-minute Walk Test, modified Activities-specific Balance Confidence Scale and SARA scale. 10 participants will complete the training program. They will be evaluated at baseline, at week 4 (miway) and after the program.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed ARSACS diagnosis; walker (indoor walking abilities with or without walking aids); ability to walk 10 meters; ability to provide informed consent

Exclusion Criteria:

* Having other medical diagnosis causing physical limitations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Change in the Scale for the assessement and rating of ataxia (SARA) | Baseline, week 4, week 8
  Measured with the Scale for the assessement and rating of ataxia (SARA), score range 0-40, higher score indicates higer ataxia severity

SECONDARY OUTCOMES:
Change in walking speed | Baseline, week 4, week 8
  Change in the walking speed, measured with the time to walk 10 meters at comfortable and maximum speed
Change in the number of sit-to-stand performed in 30 seconds | Baseline, week 4, week 8
  Number of complete sit-to-stand performed in 30 seconds without the help of arms
Change in the balance confidence | Baseline, week 4, week 8
  Measured with the modified Activities-specific Balance Confidence (ABC) Scale, score range 0-100, 0 indicates no confidence and 100 is full confidence.
Change in balance | Baseline, week 4, week 8
  Measured with the Berg Balance Scale, score range 0-56, a higher score indicates better balance.
Change in sitting balance | Baseline, week 4, week 8
  Measured with the Ottawa sitting scale, score range 0-40, a higher score indicates a better outcome.
Change in the level of independence to perform daily living activities | Baseline, week 4, week 8
  Measured with the Barthel Index, score range 0-100, a higher score indicates a higher level of independence.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gagnon, PhD, Principal Investigator — Sherbrooke University
Locations (1):
- Groupe de recherche interdisciplinaire sur les maladies neuromusculaires, Saguenay, Quebec, Canada